CLINICAL TRIAL: NCT03668119
Title: A Randomized, Open-Label, Phase 2 Study of Nivolumab in Combination With Ipilimumab or Nivolumab Monotherapy in Participants With Advanced or Metastatic Solid Tumors of High Tumor Mutational Burden (TMB-H)
Brief Title: A Study of Nivolumab Combined With Ipilimumab and Nivolumab Alone in Patients With Advanced or Metastatic Solid Tumors of High Tumor Mutational Burden (TMB-H)
Acronym: CheckMate 848
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-848; 2016-002898-35 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Pan Tumor
Keywords: TMB-H
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Ipilimumab Combination (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab Monotherapy (Experimental)
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Nivolumab + Ipilimumab Combination

SUMMARY:
The purpose of this study is to demonstrate the clinical activity of nivolumab in combination with ipilimumab in multiple types of tumors based on their Tumor Mutational Burden status.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a refractory, metastatic, or unresectable histologically or cytologically confirmed solid malignant tumor with high tumor mutational burden (TMB-H) who are refractory to standard local therapies, or for which no standard treatment is available.
* Must be able to provide tissue and blood TMB-H testing results
* Must have measurable disease for response assessment

Exclusion Criteria:

* Participants with melanoma, non-small cell lung cancer (NSCLC), renal cell carcinoma (RCC) or hematological malignancy as primary site of disease
* Participants who received prior treatment with an anti-programmed death-1 (anti-PD-1), anti-programmed death ligand 1 (anti-PD-L1), anti-programmed death ligand 2 (anti-PD-L2), anti-CD137, or anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Treatment with any chemotherapy, radiation therapy, biologics for cancer, or investigational therapy within 28 days of first administration of study treatment

Other protocol defined inclusion/exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (10):
  - John Wayne Cancer Center, Santa Monica, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Local Institution - 0093, Minneapolis, Minnesota
  - Broome Oncology, Johnson City, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Local Institution - 0079, Portland, Oregon
  - Local Institution - 0095, Austin, Texas
  - Local Institution - 0094, Dallas, Texas
  - Local Institution - 0090, Houston, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
- Argentina (5):
  - Local Institution - 0016, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Local Institution - 0087, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0078, CABA
  - Local Institution - 0015, CABA
  - Local Institution - 0119, Córdoba
- Australia (3):
  - Local Institution - 0118, St Leonards, New South Wales
  - Local Institution - 0062, Sydney, New South Wales
  - Local Institution - 0117, Woolloongabba, Queensland
- Belgium (3):
  - Local Institution - 0112, Brussels
  - Local Institution - 0113, Brussels
  - Local Institution - 0114, Leuven
- Canada (4):
  - Local Institution - 0010, Edmonton, Alberta
  - Local Institution - 0060, Hamilton, Ontario
  - Local Institution - 0036, Montreal, Quebec
  - Local Institution - 0088, Montreal, Quebec
- Chile (2):
  - Local Institution - 0018, Santiago, Santiago Metropolitan
  - Local Institution - 0082, Santiago, Santiago Metropolitan
- Denmark (2):
  - Local Institution - 0080, Copenhagen
  - Local Institution - 0081, Herlev
- France (5):
  - Local Institution - 0072, Lyon
  - Local Institution - 0075, Marseille
  - Local Institution - 0073, Paris
  - Local Institution - 0074, Toulouse
  - Local Institution - 0085, Villejuif
- Germany (5):
  - Local Institution - 0039, Berlin
  - Local Institution - 0001, Bonn
  - Local Institution - 0002, Dresden
  - Local Institution - 0086, Essen
  - Local Institution - 0043, Würzburg
- Italy (4):
  - Local Institution - 0032, Genova
  - IRCCS Istituto Nazionale Tumori Milano, Milan
  - Local Institution - 0029, Napoli
  - Local Institution - 0031, Siena
- Netherlands (2):
  - Local Institution - 0116, Rotterdam, South Holland
  - Local Institution - 0115, Amsterdam
- Poland (2):
  - Local Institution - 0076, Warsaw, Masovian Voivodeship
  - Local Institution - 0077, Gdansk
- Fundacion De Investigacion, San Juan, Puerto Rico
- Romania (5):
  - Local Institution - 0068, Cluj-Napoca, Cluj
  - Local Institution - 0069, Bucharest
  - Local Institution - 0067, Craiova
  - Local Institution - 0070, Floreşti
  - Local Institution - 0071, Timisoara, Timis
- Singapore (2):
  - Local Institution - 0065, Singapore, Central Singapore
  - Local Institution - 0066, Singapore
- Spain (3):
  - Local Institution - 0084, Barcelona
  - Local Institution - 0083, Madrid
  - Local Institution - 0110, Pamplona
- United Kingdom (2):
  - Local Institution - 0106, London, Greater London
  - Local Institution - 0107, Preston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schenker M, Burotto M, Richardet M, Ciuleanu TE, Goncalves A, Steeghs N, Schoffski P, Ascierto PA, Maio M, Lugowska I, Lupinacci L, Leary A, Delord JP, Grasselli J, Tan DSP, Friedmann J, Vuky J, Tschaika M, Konduru S, Vemula SV, Slepetis R, Kollia G, Pacius M, Duong Q, Huang N, Doshi P, Baden J, Di Nicola M. Randomized, open-label, phase 2 study of nivolumab plus ipilimumab or nivolumab monotherapy in patients with advanced or metastatic solid tumors of high tumor mutational burden. J Immunother Cancer. 2024 Aug 6;12(8):e008872. doi: 10.1136/jitc-2024-008872. PMID 39107131
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Salvage setting describes participants with a refractory, metastatic, or unresectable histologically or cytologically confirmed solid malignant tumor with Tumor Mutational Burden-High (TMB-H) who are refractory to standard therapies per local management guidelines, or for which no standard treatment per local management guidelines is available.
  Participants randomized to the Nivolumab monotherapy arm B were allowed to rollover to Nivolumab+Ipilimumab arm A at the time of progression.
Groups:
- Arm A: Nivolumab+Ipilimumab: Nivolumab 240 mg every 2 weeks (Q2W) + Ipilimumab 1 mg/kg every 6 weeks (Q6W) up to 24 months
- Arm B: Nivolumab: Nivolumab Monotherapy 480 mg every 4 weeks (Q4W) up to 24 months
Period: Pre-treatment
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Started (Randomized) | 136 | 76
bTMB-H Started (Randomized in a salvage setting) | 80 | 45
tTMB-H Started (Randomized in a salvage setting) | 88 | 47
Completed (Treated) | 135 | 76
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0
Period: Treatment
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Started (Treated) | 135 | 76
bTMB-H Started (Treated) | 83 | 47
tTMB-H Started (Treated) | 94 | 50
Arm B Rollover | 0 | 22
Completed (Continuing in the treatment period) | 0 | 0
Not Completed | 135 | 76
Not completed — Disease Progression | 76 | 57
Not completed — Study drug toxicity | 19 | 1
Not completed — Death | 3 | 0
Not completed — Adverse Event unrelated to Study drug | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Participant request to discontinue study treatment | 3 | 1
Not completed — Maximum Clinical Benefit | 0 | 1
Not completed — Participants completed treatment | 27 | 11
Not completed — Other reasons | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab | Total
Number analyzed (Participants) | 136 | 76 | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (11.7) | 57.6 (12.1) | 59.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 44 | 115
  Male | 65 | 32 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 45 | 20 | 65
  Unknown or Not Reported | 78 | 51 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 124 | 60 | 184
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR) - Arm A
Description: ORR was defined as the percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR) based on Blinded Independent Central Review (BICR) assessment.
  RECIST Criteria:
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR= ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  RANO Criteria:
  CR= Disappearance of all enhancing measurable and nonmeasurable disease; stable or improved nonenhancing T2/FLAIR lesions; off corticosteroids; and stable or improved clinically PR= ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions; no progression of nonmeasureable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; and stable or improved clinically.
Time Frame: From date of randomization up to 42 months
Population: All participants randomized in a salvage setting to arm A by TMB-High status
Measure: Number (95% Confidence Interval); unit: Precentage of participants
Arm/Group | Arm A: Nivolumab+Ipilimumab
Number analyzed (Participants) | 88
Precentage of participants
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80
  Blood TMB-H (bTMB-H) | 22.5 [13.9 to 33.2]
  Tissue TMB-H (tTMB-H) | 38.6 [28.4 to 49.6]

2. Secondary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR) - Arm B
Description: as for outcome 1
Time Frame: From date of randomization up to 57 months
Population: All participants randomized in a salvage setting to arm B by TMB-High status
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm B: Nivolumab
Number analyzed (Participants) | 47
Percentage of participants
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 45
  Blood TMB-H (bTMB-H) | 15.6 [6.5 to 29.5]
  Tissue TMB-H (tTMB-H) | 29.8 [17.3 to 44.9]

3. Secondary Outcome: Objective Response Rate (ORR) Per Investigator
Description: ORR was defined as the percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR) based on investigator assessment. Calculated using Clopper-Pearson method.
  RECIST Criteria:
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR= ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  RANO Criteria:
  CR= Disappearance of all enhancing measurable and nonmeasurable disease; stable or improved nonenhancing T2/FLAIR lesions; off corticosteroids; and stable or improved clinically PR= ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions; no progression of nonmeasureable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; and stable or improved clinically.
Time Frame: From date of randomization up to 57 months
Population: All participants randomized in a salvage setting by TMB-High status
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 88 | 47
Percentage of participants
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80 | 45
  Blood TMB-H (bTMB-H) | 25.0 [16.0 to 35.9] | 13.3 [5.1 to 26.8]
  Tissue TMB-H (tTMB-H) | 44.3 [33.7 to 55.3] | 23.4 [12.3 to 38.0]

4. Secondary Outcome: Duration of Response (DoR) Per Investigator
Description: DoR was defined as the time from first confirmed complete or partial response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first. Calculated using KM method.
  RECIST Criteria:
  CR= Disappearance of all target lesions. PR= ≥ 30% decrease in the sum of diameters of target lesions. PD= ≥ 20% increase in the sum of diameters of target lesions.
  RANO Criteria:
  CR= Disappearance of all enhancing measurable and nonmeasurable disease; stable/improved T2/FLAIR; off corticosteroids; stable/improved clinically PR= ≥ 50% decrease in the sum of diameters of all measurable enhancing lesions; no progression of nonmeasurable disease; no new lesions; stable/improved T2/FLAIR; stable/improved clinically.
  PD= ≥ 25% increase in sum of diameters of enhancing lesions, on stable/increasing doses of corticosteroids; significant increase in T2/FLAIR; any new lesion; clear clinical deterioration or clear progression of nonmeasurable disease.
Time Frame: From date of randomization to date of first documented tumor progression, or date of death, whichever occurs first (Up to 57 months)
Population: All responders (CR or PR) randomized in a salvage setting by TMB-High status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 39 | 11
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 20 | 6
  Blood TMB-H (bTMB-H) | 27.96 [11.20 to NA] — insufficient number of participants with events | NA [11.24 to NA] — insufficient number of participants with events
  Tissue TMB-H (tTMB-H) | NA [27.96 to NA] — insufficient number of participants with events | NA [8.05 to NA] — insufficient number of participants with events

5. Secondary Outcome: Duration of Response (DoR) Per Blinded Independent Central Review (BICR)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All responders (CR or PR) randomized in a salvage setting by TMB-High status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 34 | 14
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 18 | 7
  Blood TMB-H (bTMB-H) | NA [10.15 to NA] — insufficient number of participants with events | NA [5.52 to NA] — insufficient number of participants with events
  Tissue TMB-H (tTMB-H) | NA [33.51 to NA] — insufficient number of participants with events | NA [8.31 to NA] — insufficient number of participants with events

6. Secondary Outcome: Time to Objective Response (TTR) Per Investigator
Description: TTR is defined as the time from randomization date to the date of the first confirmed response (complete response (CR) or partial response (PR)), based on investigator assessment.
  RECIST Criteria:
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR= ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  RANO Criteria:
  CR= Disappearance of all enhancing measurable and nonmeasurable disease; stable or improved nonenhancing T2/FLAIR lesions; off corticosteroids; and stable or improved clinically PR= ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions; no progression of nonmeasureable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; and stable or improved clinically.
Time Frame: From date of randomization to date of first confirmed response (CR or PR) (Up to 57 months)
Population: All responders (CR or PR) randomized in a salvage setting by TMB-High status
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 39 | 11
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 20 | 6
  Blood TMB-H (bTMB-H) | 3.48 (1.17) | 4.08 (3.40)
  Tissue TMB-H (tTMB-H) | 3.56 (1.74) | 3.75 (2.50)

7. Secondary Outcome: Time to Objective Response (TTR) Per Blinded Independent Central Review (BICR)
Description: TTR is defined as the time from randomization date to the date of the first confirmed response (complete response (CR) or partial response (PR)), based on Blinded Independent Central Review (BICR) assessment.
  RECIST Criteria:
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR= ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  RANO Criteria:
  CR= Disappearance of all enhancing measurable and nonmeasurable disease; stable or improved nonenhancing T2/FLAIR lesions; off corticosteroids; and stable or improved clinically PR= ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions; no progression of nonmeasureable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; and stable or improved clinically.
Time Frame: From date of randomization to date of first confirmed response (CR or PR) (Up to 57 months)
Population: All responders (CR or PR) randomized in a salvage setting by TMB-High status
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 34 | 14
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 18 | 7
  Blood TMB-H (bTMB-H) | 3.59 (1.65) | 4.33 (2.93)
  Tissue TMB-H (tTMB-H) | 4.37 (5.10) | 3.98 (2.47)

8. Secondary Outcome: Clinical Benefit Rate (CBR) Per Investigator
Description: CBR is defined as the percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR) or stable disease (SD) based on investigator assessment.
  RECIST Criteria:
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm PR= ≥ 30% decrease in the sum of diameters of target lesions SD= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
  RANO Criteria:
  CR= Disappearance of all enhancing disease; stable or improved nonenhancing T2/FLAIR lesions; off corticosteroids; and stable or improved clinically PR= ≥ 50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions; no progression of nonmeasureable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions; stable or improved clinically SD= does not qualify for CR, PR, or progression; stable nonenhancing T2/FLAIR lesions
Time Frame: From date of randomization up to 57 months
Population: All participants randomized in a salvage setting by TMB-High status
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 88 | 47
Percentage of participants
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80 | 45
  Blood TMB-H (bTMB-H) | 42.5 [31.5 to 54.1] | 40.0 [25.7 to 55.7]
  Tissue TMB-H (tTMB-H) | 63.6 [52.7 to 73.6] | 46.8 [32.1 to 61.9]

9. Secondary Outcome: Clinical Benefit Rate (CBR) Per Blinded Independent Central Review (BICR)
Description: CBR is defined as the percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR) or stable disease (SD) per Blinded Independent Central Review (BICR) assessment.
  RECIST Criteria:
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm PR= ≥ 30% decrease in the sum of diameters of target lesions SD= does not qualify for PR or progressive disease
  RANO Criteria:
  CR= Disappearance of all enhancing disease; stable or improved nonenhancing T2/FLAIR lesions; off corticosteroids; and stable or improved clinically PR= ≥ 50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions; no progression of nonmeasureable disease; no new lesions; stable or improved nonenhancing (T2/FLAIR) lesions; stable or improved clinically SD= does not qualify for CR, PR, or progression; stable nonenhancing T2/FLAIR lesions
Time Frame: From date of randomization up to 57 months
Population: All participants randomized in a salvage setting by TMB-High status
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 88 | 47
Percentage of participants
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80 | 45
  Blood TMB-H (bTMB-H) | 32.5 [22.4 to 43.9] | 28.9 [16.4 to 44.3]
  Tissue TMB-H (tTMB-H) | 53.4 [42.5 to 64.1] | 38.3 [24.5 to 53.6]

10. Secondary Outcome: Progression Free Survival (PFS) Per Investigator
Description: PFS is defined as the time from randomization date to the date of the first documented tumor progression, determined by investigator assessment, or death due to any cause, whichever occurs first. Calculated using KM method.
  RECIST Criteria:
  Progressive Disease (PD)= ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of ≥ 5 mm.
  RANO Criteria:
  PD= ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline or best response, on stable or increasing doses of corticosteroids; significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy; any new lesion; clear clinical deterioration or clear progression of nonmeasurable disease.
Time Frame: as for outcome 4
Population: All participants randomized in a salvage setting by TMB-High status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 88 | 47
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80 | 45
  Blood TMB-H (bTMB-H) | 2.99 [2.66 to 4.34] | 3.04 [2.79 to 5.36]
  Tissue TMB-H (tTMB-H) | 8.15 [4.83 to 12.94] | 3.06 [2.79 to 10.91]

11. Secondary Outcome: Progression Free Survival (PFS) Per Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from randomization date to the date of the first documented tumor progression, determined by Blinded Independent Central Review (BICR) assessment, or death due to any cause, whichever occurs first. Calculated using KM method.
  RECIST Criteria:
  Progressive Disease (PD)= ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of ≥ 5 mm.
  RANO Criteria:
  PD= ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline or best response, on stable or increasing doses of corticosteroids; significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy; any new lesion; clear clinical deterioration or clear progression of nonmeasurable disease.
Time Frame: as for outcome 4
Population: All participants randomized in a salvage setting by TMB-High status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 88 | 47
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80 | 45
  Blood TMB-H (bTMB-H) | 2.83 [2.33 to 2.99] | 2.83 [2.60 to 3.25]
  Tissue TMB-H (tTMB-H) | 5.68 [3.19 to 11.60] | 2.83 [2.69 to 5.72]

12. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death due to any cause. Participants who did not have a date of death were censored on the last date for which a participant was known to be alive. Calculated using KM method.
Time Frame: From date of randomization to date of death (Up to 57 months)
Population: All participants randomized in a salvage setting by TMB-High status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 88 | 47
Months
  Blood TMB-H (bTMB-H): number analyzed (Participants) | 80 | 45
  Blood TMB-H (bTMB-H) | 8.07 [5.82 to 10.45] | 11.24 [5.26 to 18.99]
  Tissue TMB-H (tTMB-H) | 16.48 [10.18 to 30.52] | 14.59 [7.69 to 18.23]

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with any grade adverse events (AEs), serious adverse events (SAEs), drug-related AEs, and drug-related SAEs by Tumor Mutational Burden- High (TMB-H) status using worst grade per national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) v5 criteria. An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  TMB-H = ≥ 10 mutations per megabase bTMB-H and tTMB-H are not mutually exclusive
Time Frame: From first dose to 30 days post last dose (Up to 25 months)
Population: All treated participants by TMB-High status
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 94 | 50
Participants
  Blood TMB-H (bTMB-H) AEs: number analyzed (Participants) | 83 | 47
  Blood TMB-H (bTMB-H) AEs | 82 | 46
  Tissue TMB-H (tTMB-H) AEs | 93 | 50
  bTMB-H SAEs: number analyzed (Participants) | 83 | 47
  bTMB-H SAEs | 51 | 17
  tTMB-H SAEs | 46 | 16
  bTMB-H drug-related AEs: number analyzed (Participants) | 83 | 47
  bTMB-H drug-related AEs | 64 | 29
  tTMB-H drug-related AEs | 78 | 27
  bTMB-H drug-related SAEs: number analyzed (Participants) | 83 | 47
  bTMB-H drug-related SAEs | 17 | 1
  tTMB-H drug-related SAEs | 16 | 2

14. Secondary Outcome: Number of Participants With On-Treatment Laboratory Parameters
Description: Number of participants with grade 3-4 on-treatment laboratory parameters. Parameters include hematology, chemistry, liver function, and renal function using worst grade per national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) v5 criteria.
  Grade 3=Severe event Grade 4=Life threatening event TMB-H = ≥ 10 mutations per megabase bTMB-H and tTMB-H are not mutually exclusive
Time Frame: From first dose to 30 days post last dose (Up to 25 months)
Population: All treated participants with on-treatment laboratory measures by TMB-H status
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab
Number analyzed (Participants) | 91 | 45
Participants
  Blood TMB-H (bTMB-H) Hemoglobin grade 3: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Hemoglobin grade 3 | 6 | 3
  Tissue TMB-H (tTMB-H) Hemoglobin grade 3 | 8 | 7
  Blood TMB-H (bTMB-H) Platelet Count grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Platelet Count grade 3-4 | 1 | 0
  Tissue TMB-H (tTMB-H) Platelet Count grade 3-4 | 0 | 1
  Blood TMB-H (bTMB-H) Leukocytes grade 3- 4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Leukocytes grade 3- 4 | 1 | 0
  Tissue TMB-H (tTMB-H) Leukocytes grade 3- 4 | 0 | 0
  Blood TMB-H (bTMB-H) Leukocytes Absolute grade 3- 4: number analyzed (Participants) | 70 | 39
  Blood TMB-H (bTMB-H) Leukocytes Absolute grade 3- 4 | 2 | 1
  Tissue TMB-H (tTMB-H) Leukocytes Absolute grade 3- 4: number analyzed (Participants) | 76 | 40
  Tissue TMB-H (tTMB-H) Leukocytes Absolute grade 3- 4 | 5 | 3
  Blood TMB-H (bTMB-H) Absolute Neutrophil grade 3- 4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Absolute Neutrophil grade 3- 4 | 1 | 1
  Tissue TMB-H (tTMB-H) Absolute Neutrophil grade 3- 4 | 0 | 0
  Blood TMB-H (bTMB-H) Alkaline Phosphatase grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Alkaline Phosphatase grade 3-4 | 2 | 1
  Tissue TMB-H (tTMB-H) Alkaline Phosphatase grade 3-4 | 2 | 0
  Blood TMB-H (bTMB-H) Aspartate Aminotransferase grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Aspartate Aminotransferase grade 3-4 | 2 | 3
  Tissue TMB-H (tTMB-H) Aspartate Aminotransferase grade 3-4 | 4 | 1
  Blood TMB-H (bTMB-H) Alanine Aminotransferase grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Alanine Aminotransferase grade 3-4 | 5 | 2
  Tissue TMB-H (tTMB-H) Alanine Aminotransferase grade 3-4 | 3 | 1
  Blood TMB-H (bTMB-H) Bilirubin grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Bilirubin grade 3-4 | 3 | 2
  Tissue TMB-H (tTMB-H) Bilirubin grade 3-4 | 3 | 1
  Blood TMB-H (bTMB-H) Creatinine grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Creatinine grade 3-4 | 3 | 1
  Tissue TMB-H (tTMB-H) Creatinine grade 3-4 | 3 | 0
  Blood TMB-H (bTMB-H) Hypernatremia grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Hypernatremia grade 3-4 | 0 | 0
  Tissue TMB-H (tTMB-H) Hypernatremia grade 3-4 | 0 | 0
  Blood TMB-H (bTMB-H) Hyponatremia grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Hyponatremia grade 3-4 | 4 | 1
  Tissue TMB-H (tTMB-H) Hyponatremia grade 3-4 | 3 | 1
  Blood TMB-H (bTMB-H) Hyperkalemia grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Hyperkalemia grade 3-4 | 2 | 0
  Tissue TMB-H (tTMB-H) Hyperkalemia grade 3-4 | 2 | 0
  Blood TMB-H (bTMB-H) Hypokalemia grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Hypokalemia grade 3-4 | 4 | 0
  Tissue TMB-H (tTMB-H) Hypokalemia grade 3-4 | 3 | 1
  Blood TMB-H (bTMB-H) Hypercalcemia grade 3-4: number analyzed (Participants) | 77 | 43
  Blood TMB-H (bTMB-H) Hypercalcemia grade 3-4 | 0 | 1
  Tissue TMB-H (tTMB-H) Hypercalcemia grade 3-4 | 2 | 0
  Blood TMB-H (bTMB-H) Hypocalcemia grade 3-4: number analyzed (Participants) | 77 | 43
  Blood TMB-H (bTMB-H) Hypocalcemia grade 3-4 | 2 | 0
  Tissue TMB-H (tTMB-H) Hypocalcemia grade 3-4 | 0 | 1
  Blood TMB-H (bTMB-H) Hyperglycemia grade 3-4: number analyzed (Participants) | 39 | 26
  Blood TMB-H (bTMB-H) Hyperglycemia grade 3-4 | 0 | 0
  Tissue TMB-H (tTMB-H) Hyperglycemia grade 3-4: number analyzed (Participants) | 52 | 26
  Tissue TMB-H (tTMB-H) Hyperglycemia grade 3-4 | 0 | 0
  Blood TMB-H (bTMB-H) Hypoglycemia grade 3-4: number analyzed (Participants) | 77 | 44
  Blood TMB-H (bTMB-H) Hypoglycemia grade 3-4 | 0 | 0
  Tissue TMB-H (tTMB-H) Hypoglycemia grade 3-4 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and AEs are assessed from first dose to 100 days post last dose (Up to 27 months). Participants were assessed for all-cause mortality from their first dose to study completion (Up to 57 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Arm B: Nivolumab+Ipilimumab (Rollover): Nivolumab 240 mg every 2 weeks (Q2W) + Ipilimumab 1 mg/kg every 6 weeks (Q6W)
Arm/Group | Arm A: Nivolumab+Ipilimumab | Arm B: Nivolumab | Arm B: Nivolumab+Ipilimumab (Rollover)
All-Cause Mortality (participants affected / at risk) | 97/136 | 42/76 | 20/22
Serious Adverse Events (participants affected / at risk) | 90/135 | 39/76 | 11/22
Other Adverse Events (participants affected / at risk) | 121/135 | 64/76 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab+Ipilimumab (N=135) | Arm B: Nivolumab (N=76) | Arm B: Nivolumab+Ipilimumab (Rollover) (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Pericarditis malignant (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 2 | 0 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 4 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Death (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 0
General physical health deterioration (General disorders) | 2 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0
Prostate infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 1
Urosepsis (Infections and infestations) | 2 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary tract injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 43 | 25 | 7
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Obstructive nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine fistula (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab+Ipilimumab (N=135) | Arm B: Nivolumab (N=76) | Arm B: Nivolumab+Ipilimumab (Rollover) (N=22)
Anaemia (Blood and lymphatic system disorders) | 32 | 16 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 5 | 0
Hyperthyroidism (Endocrine disorders) | 15 | 3 | 1
Hypothyroidism (Endocrine disorders) | 18 | 11 | 0
Abdominal pain (Gastrointestinal disorders) | 23 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 23 | 10 | 1
Diarrhoea (Gastrointestinal disorders) | 50 | 14 | 3
Dry mouth (Gastrointestinal disorders) | 6 | 6 | 0
Nausea (Gastrointestinal disorders) | 19 | 15 | 4
Vomiting (Gastrointestinal disorders) | 19 | 7 | 3
Asthenia (General disorders) | 16 | 10 | 1
Fatigue (General disorders) | 41 | 17 | 2
Oedema peripheral (General disorders) | 22 | 5 | 0
Pyrexia (General disorders) | 21 | 10 | 2
COVID-19 (Infections and infestations) | 10 | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 12 | 2 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 4 | 0
Alanine aminotransferase increased (Investigations) | 19 | 8 | 2
Amylase increased (Investigations) | 7 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 20 | 12 | 1
Blood alkaline phosphatase increased (Investigations) | 13 | 8 | 1
Blood bilirubin increased (Investigations) | 10 | 7 | 0
Blood creatinine increased (Investigations) | 11 | 7 | 2
Blood glucose increased (Investigations) | 7 | 3 | 0
Weight decreased (Investigations) | 4 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 28 | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0
Headache (Nervous system disorders) | 11 | 4 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 4 | 0
Insomnia (Psychiatric disorders) | 13 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 15 | 8
Rash (Skin and subcutaneous tissue disorders) | 25 | 7 | 1
Hypotension (Vascular disorders) | 7 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03668119/Prot_SAP_000.pdf